CLINICAL TRIAL: NCT03546556
Title: 18-FLT PET/MR Imaging to Predict Graft Failure and Graft Versus Host Disease in Bone Marrow Transplant Patients
Brief Title: 18-FLT PET/MR Imaging to Predict Graft Failure and GVHD in Bone Marrow Transplant Patients
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study terminated due to COVID-19 pandemic and not being able to perform PET/MR scans on participants.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC 1714
Record Dates: First submitted 2018-03-19; First posted 2018-06-06 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Graft Vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — alovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Allogeneic (Experimental): A total of 12 patients who have undergone allogenic bone marrow transplantation will undergo Fluorothymidine FLT-PET-MRI imaging on two separate occasions.
  Interventions: Drug: Fluorothymidine (FLT)
- Autologous (Experimental): 3 patients undergoing autologous stem cell transplant will also undergo Fluorothymidine FLT-PET-MRI imaging the same two time points in order to determine how much of the FLT signal observed after allogeneic transplant is unique to that population and the result of allo-antigen driven T cell expansion.
  Interventions: Drug: Fluorothymidine (FLT)

INTERVENTIONS:
Drug: Fluorothymidine (FLT) — A total of 12 patients who have undergone allogenic bone marrow transplantation will undergo FLT-PET-MRI imaging on two separate occasions. In addition to the 12 allogenic transplant patients, 3 patients undergoing autologous stem cell transplant will also be imaged the same two time points in order to determine how much of the FLT signal observed after allogeneic transplant is unique to that population and the result of allo-antigen driven T cell expansion.
  Other Names: 18F-FLT; 3'-deoxy-3'-(18F) fluorothymidine; 3'-deoxy-3'-[18F]fluorothymidine; fluorothymidine F 18; fluorothymidine F-18; Thymidine, 3'-deoxy-3'-(18F)fluoro-

SUMMARY:
Allogeneic HSCT is potentially curative for numerous high risk hematologic malignancies and offers several advantages over traditional chemotherapy. First, higher doses of cytotoxic chemotherapy and/or irradiation can be given since patients are subsequently rescued from the severe myelosuppression induced by the pre-transplant conditioning regimen by the infusion of healthy hematopoietic stem cells.

Second and perhaps more importantly, mature T cells contained in the graft are able to mount immune responses against residual cancer cells surviving the conditioning regimen due to major and/or minor MHC disparities between the donor and recipient. Unfortunately, the allo-immune responses driving the GVL effect are typically not specific for malignant cells. As a consequence, donor immune cells attack normal host tissues resulting in a process known as acute graft-versus-host disease (GVHD). Acute GVHD is primarily T cell driven, usually occurs within the first few months after transplant, and results in skin rash, diarrhea, cholestatic liver damage, and, on occasion, acute lung injury.

DETAILED DESCRIPTION:
The current proposal explores the use of a novel imaging modality, FLT PET/MRI, to correlate allogeneic transplant outcomes with FLT and MRI findings during early stem cell engraftment and at a later time point following stable count recovery. Specifically, this study will determine if the strength of the early FLT signal within the bone marrow correlates with engraftment success and if isolated areas of cellular proliferation within the marrow at a later time point might predict for leukemia relapse. In addition, based on the important role that host lymphoid tissues are known to play in GVHD pathogenesis in mice, this study will determine if the FLT signal within host SLT after transplant can predict for the development of GVHD in human BMT patients. Because FLT imaging by itself cannot distinguish between bone marrow engraftment/proliferation and the allo-immune driven T cell expansion that ultimately results in GVHD, this study will image autologous transplant patients as a comparator arm. Autologous HSCT like allogeneic transplantation involves the administration of very high doses of chemotherapy to high risk cancer patients in order to achieve better tumor kill. However, in this situation patients are administered their own cryopreserved stem cells to reconstitute the ablated hematopoietic system. Under those circumstances there is no allo-immune reactivity to drive T cell activation and expansion after transplant, and as a result there is no GVHD in the autologous transplant setting. Thus, these patients will help us to elucidate how much of the FLT signal seen in the allogeneic setting is the result of allo-immune driven T cell expansion.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing allogeneic bone marrow transplant for acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), or myelodysplastic syndrome
* Allogeneic transplant patients receiving either a fully myeloablative or reduced intensity chemotherapy +/- total body irradiation (TBI) conditioning regimen are eligible.
* Allogeneic transplant patients receiving stem cells from a matched related, matched unrelated, mismatched unrelated, mismatched related (including haplotype matched) donors are eligible
* Allogeneic transplant patients must be in a complete morphologic remission prior to transplant
* Patients undergoing autologous bone marrow transplant for multiple myeloma
* Myeloma patients must have achieved at least a very good partial remission prior to transplant and exhibit fewer than 10% plasma cells in their pre-transplant marrow biopsy
* At least 18 years of age
* Negative urine pregnancy test in women of child-bearing potential

Exclusion Criteria:

* Any woman who is pregnant or has reason to believe she is pregnant or any woman who is lactating.
* Condition that makes MRI unsafe (e.g., cardiac pacemaker, epicardial pacemaker leads, cochlear implants, metal aneurysm clip, metal halo devices)
* Inability to tolerate MRI (e.g., unable to lie flat for > 1 hour, severe claustrophobia)
* Known allergy to fluorothymidine
* Creatinine clearance < 40 ml/min, as estimated by the Cockcroft-Gault formula
* Body Mass Index (BMI) > 35
* Poorly controlled diabetes mellitus (fasting blood glucose > 500 mg/dl)
* Institutionalized subject (prisoner or nursing home patient)
* Critically ill or medically unstable
* Currently hospitalized (All FLT PET/MR scans will be obtained in the outpatient setting)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Overall FLT-PET Bone Marrow Signal | 35 Days (Approximate)
  Compare the overall FLT-PET bone marrow signal on transplant day +25 between allogeneic stem cell transplant recipients who do and do not go on to achieve complete donor bone marrow reconstitution by transplant day +35.
Overall FLT-PET Signal Intensity within Host Secondary Lymphoid Sites | 100 Days (Approximate)
  Compare the overall FLT-PET signal intensity within host secondary lymphoid sites on transplant day +60 between allogeneic stem cell transplant recipients who do and do not develop acute GVHD by transplant day +100.

SECONDARY OUTCOMES:
Overall Long-Term FLT-PET Bone Marrow Signal | 100 Days (Approximate)
  Compare the overall FLT-PET bone marrow signal on transplant day +60 between allogeneic stem cell transplant recipients who do and do not achieve complete donor bone marrow reconstitution by transplant day +100.
Overall Long-Term FLT-PET Signal Intensity within Host Secondary Lymphoid Sites | 100 Days (Approximate)
  Compare the overall FLT-PET signal intensity within host secondary lymphoid sites on transplant day +25 between allogeneic stem cell transplant recipients who do and do not develop acute GVHD by transplant day +100.
Differences in FLT Uptake in Autologous HSCT and Allogeneic HSCT Patients | 100 Days (Approximate)
  Evaluate differences in FLT uptake within the bone marrow and secondary lymphoid tissues in patients undergoing autologous hematopoietic stem cell transplantation (HSCT) versus allogeneic HSCT.
Strength of FLT-PET Signal and Transfusion Independence | 35 Days (Approximate)
  Correlate the strength of the FLT-PET signal within the bone marrow on transplant day +25 with the rate of transfusion independence on transplant day +35 in allogeneic stem cell transplant recipients.
Strength of the FLT-PET Signal and Bone Marrow Cellularity | 35 Days (Approximate)
  Correlate the strength of the FLT-PET signal within the bone marrow on transplant day +25 with bone marrow cellularity on transplant day +35 in allogeneic stem cell transplant recipients.
Strength of FLT-PET Signal and Transfusion Independence (Long Term) | 100 Days (Approximate)
  Correlate the strength of the FLT-PET signal within the bone marrow on transplant day +60 with the rate of transfusion independence on transplant day +100 in allogeneic stem cell transplant recipients.
Strength of FLT-PET Signal and Bone Marrow Cellularity (Long Term) | 100 Days (Approximate)
  Correlate the strength of the FLT-PET signal within the bone marrow on transplant day +60 with bone marrow cellularity on transplant day +100 in allogeneic stem cell transplant recipients.
Isolated/Asymmetric Foci of Increased FLT | 100 Days (Approximate)
  Evaluate if isolated or asymmetric foci of increased FLT within the bone marrow or lymph nodes on transplant day +60 are associated with the incidence of disease relapse by day +100 in allogeneic stem cell transplant recipients.
Strength of FLT-PET signal and MRI Findings | 60 Days (Approximate)
  Correlate the strength of the FLT-PET signal within the bone marrow on transplant day +25 and on day +60 with MRI findings suggestive of engraftment in allogeneic stem cell transplant recipients.
Overall FLT-PET Signal Intensity and Acute Graft Versus Host Disease | 60 Days (Approximate)
  Evaluate the association of the overall FLT-PET signal intensity within host secondary lymphoid sites on transplant day +60 with the overall incidence of acute graft versus host disease and malignancy relapse over the first transplant year.

CONTACTS AND LOCATIONS:
Overall Officials: Z Lee, MD/PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT03546556/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT03546556/ICF_001.pdf